CLINICAL TRIAL: NCT01720511
Title: Pilot Study of the Effect of Purple Rice on Glucose Tolerance, Serum Lipids and Inflammation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PBRC 12002
Record Dates: First submitted 2012-10-30; First posted 2012-11-02 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Purple Rice (Experimental): Twice a day given purple rice with 5mg of resveratrol.
  Interventions: Dietary Supplement: Purple Rice
- Brown RIce (Active Comparator): Plain Purple rice given twice a day
  Interventions: Dietary Supplement: Brown Rice

INTERVENTIONS:
Dietary Supplement: Purple Rice — Incorporate one cup of purple rice into dishes to be consumed at lunch and dinner each day for 4 weeks (equivalent of 4 ounces of uncooked rice/day).
  Arms: Purple Rice
Dietary Supplement: Brown Rice — Incorporate one cup of brown rice into dishes to be consumed at lunch and dinner each day for 4 weeks (equivalent of 4 ounces of uncooked rice/day).
  Arms: Brown RIce

SUMMARY:
This is a pilot study to demonstrate the effect of purple rice on post-prandial glucose and insulin. The purple color is due, like red wine grapes, mainly to the anthocyanins. The safety and tolerability of purple rice is similar to white or brown rice, but contains the purple elements common to other foods like grapes.

DETAILED DESCRIPTION:
This is a study that will have 1 screening visit and 9 study visits. Subjects will come to the screening visit for blood chemistry, health questionnaire and speak to the coordinator. Each subject passing inclusion/exclusion will go on to eat purple rice for 4 weeks and brown rice for 4 weeks. The 4-week feeding periods will be balanced and assigned randomly. The subjects will report to the metabolic kitchen to pick up their supply of 14 frozen rice dishes each week in a container and return the empty containers as a measure of compliance. At the end of each 4-week feeding period, subjects will come to the inpatient unit fasting from 9pm the prior night except for water. Subjects will have an intravenous line placed and fasting blood will be drawn for chemistry. Subjects will then be given glucose to drink and blood will be drawn from then IV line for glucose and insulin at time listed in the consent.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy male or female with a fasting glucose between 100 mg/mL and 126 mg/dL or with type 2 diabetes controlled on diet without diabetes medications.
* Eighteen years of age or older.
* Hemoglobin A1c(HgbA1c) less than 7%.

Exclusion Criteria:

* Pregnant or nursing.
* Taking a medication for diabetes (e.g. Metformin), a medication known to affect blood sugar (e.g. glucocorticoids), an anti-inflammatory medication (e.g. aspiring) or triglycerides (e.g. fibrates).
* Any chronic medication that has not had a stable dose for 1 month or longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Glucose Tolerance | 10 weeks
  Subjects will have an Intravenous line placed and fasting blood will be drawn. Subjects will then be given glucose to drink and blood will be drawn from an IV line for glucose and insulin.

SECONDARY OUTCOMES:
Serum Lipids | 10 weeks
  Subjects will have an Intravenous line placed and fasting blood will be drawn for a chemistry-15 panel and High-sensitivity C-reaction Protein. Subjects will then be given 75 grams of glucose to drink and blood will be drawn from an IV line for glucose and insulin.
Inflammation measured by highly sensitive C-reative protein test | 10 weeks
  A high-sensitivity CRP (hs-CRP), that can be done in the lab using a blood test.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States